CLINICAL TRIAL: NCT02110693
Title: The TAPS Tool: Screen and Brief Assessment Tool Validation Study
Brief Title: The Tobacco, Alcohol, Prescription Medication and Other Substances Tool
Acronym: CTN0059
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Johns Hopkins University (Other); Virginia Commonwealth University (Other); NYU Langone Health (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CTN 0059; 2U10DA013034 (NIH)
Record Dates: First submitted 2014-04-02; First posted 2014-04-10 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Substance Use Disorder
Keywords: Substance Use; Substance Use Disorder; Screening; Brief Assessment
MeSH Terms: conditions — Substance-Related Disorders | interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: This study examined the accuracy of a substance abuse screening test compared to gold standard measures Participants all received the experimental screening instrument (via self- and tablet computer administration. The order of administration was randomly selected in order to control for an order effect.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interviewer and tablet administration (Other): All participants were administered the TAPS Tool via interviewer and tablet computer self-administration in the same session.
  Interventions: Other: Interviewer and tablet administration of the TAPS Tool

INTERVENTIONS:
Other: Interviewer and tablet administration of the TAPS Tool — All participant will self-administer substance use screening instrument (TAPS Tool) on a tablet computer and will be administered the TAPS Tool by an interviewer.

SUMMARY:
The purpose of the study is to develop and validate a questionnaire to screen and assess adult primary care patients for tobacco, alcohol, prescription drug, and drug use and problems related to their use.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patients
* Able to provide informed consent

Exclusion Criteria:

* inability to comprehend spoken English
* inability to self-administer the instrument on the tablet computer due to physical limitations
* previously enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2057 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Schwartz, M.D., Principal Investigator — Friends Research Institute, Inc.; Li-Tzy Wu, Psy.D., Principal Investigator — Duke University; Jennifer McNeely, M.D., Principal Investigator — New York University
Locations (4):
- United States (4):
  - Chase Brexton Health Services, Baltimore, Maryland
  - Bellevue Hospital, New York, New York
  - MURDOCK Study, Kannapolis, North Carolina
  - Virginia Commonwealth University Health System Ambulatory Care Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McNeely J, Wu LT, Subramaniam G, Sharma G, Cathers LA, Svikis D, Sleiter L, Russell L, Nordeck C, Sharma A, O'Grady KE, Bouk LB, Cushing C, King J, Wahle A, Schwartz RP. Performance of the Tobacco, Alcohol, Prescription Medication, and Other Substance Use (TAPS) Tool for Substance Use Screening in Primary Care Patients. Ann Intern Med. 2016 Nov 15;165(10):690-699. doi: 10.7326/M16-0317. Epub 2016 Sep 6. PMID 27595276
- [Derived] Wu LT, McNeely J, Subramaniam GA, Sharma G, VanVeldhuisen P, Schwartz RP. Design of the NIDA clinical trials network validation study of tobacco, alcohol, prescription medications, and substance use/misuse (TAPS) tool. Contemp Clin Trials. 2016 Sep;50:90-7. doi: 10.1016/j.cct.2016.07.013. Epub 2016 Jul 19. PMID 27444426

RESULTS

PARTICIPANT FLOW:
Groups:
- Interviewer Then Tablet Administration: Interviewer will administer the substance use screening instrument first then self-administration of the same instrument on a tablet computer
- Tablet First Then Interviewer Administration: Self-administration on tablet computer of screening instrument first, then interviewer administration of the same instrument.
Period: Overall Study
Arm/Group | Interviewer Then Tablet Administration | Tablet First Then Interviewer Administration
Started | 1026 | 1031
Completed | 998 | 1002
Not Completed | 28 | 29
Not completed — Withdrawal by Subject | 6 | 7
Not completed — skipped assessment | 15 | 18
Not completed — technical difficulties | 6 | 4
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Interviewer and Tablet Administration of TAPS Tool: All participants self-administered TAPS Tool on a computer tablet and were administered the TAPS Tool by an interviewer
Arm/Group | Interviewer and Tablet Administration of TAPS Tool
Number analyzed (Participants) | 2,000
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data (n=1) and refused to answer (n=1)
  Participants
    number analyzed (Participants) | 1,998
    Female | 1124
    Male | 874
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 233
  Not Hispanic or Latino | 1761
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participant chose not to answer (n=7)
  Participants
    American Indian or Alaska Native | 12
    Asian | 35
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1112
    White | 667
    More than one race | 66
    Unknown or Not Reported | 108
Region of Enrollment [Number; unit: participants]
  United States | 2000

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic and Statistical Manual-5 (DSM-5) Alcohol Use Disorder Diagnosis Measured by the Modified World Mental Health Composite International Diagnostic Interview
Description: The Modified World Mental Health Composite International Diagnostic Interview is a structured interview that assesses whether or not the participant meets DSM-5 Diagnostic Criteria
Time Frame: Baseline
Population: Adult primary care patients
Measure: Number (95% Confidence Interval); unit: Sensitivity
Groups:
- Interviewer Administration: Interviewer administration of a substance misuse screening instrument (TAPS Tool).
- Tablet Administration: Self-administration on tablet computer of screening instrument for substance misuse (TAPS Tool).
Arm/Group | Interviewer Administration | Tablet Administration
Number analyzed (Participants) | 2000 | 2000
Sensitivity | .70 [.64 to .75] | .74 [.68 to .79]
Statistical Analysis 1: Comparison: Interviewer Administration; Each administration approach (interviewer and tablet) was tested separately against the reference measure; Test type: Other — Concurrent validity of the interviewer and self-administered versions of the TAPS Tool compared to the reference standard was assessed for Alcohol Use Disorder using receiver operator characteristic (ROC) curves; Sensitivity = .70, 95% CI 2-sided [.64 to .75]
Statistical Analysis 2: Comparison: Tablet Administration; Each administration approach (interviewer and tablet) was tested separately against the reference measure; Test type: Other — [test comment as in outcome 1, analysis 1]; Sensitivity = .74, 95% CI 2-sided [.68 to .79]

2. Primary Outcome: Diagnostic and Statistical Manual-5 (DSM-5) Cannabis Use Disorder Diagnosis Measured With Modified World Mental Health Composite International Diagnostic Interview
Description: as for outcome 1
Time Frame: Baseline
Population: Adult primary care population
Measure: Number (95% Confidence Interval); unit: Sensitivity
Groups:
- Tablet Administration: Tablet computer administration of a substance misuse screening instrument (TAPS Tool).
Arm/Group | Interviewer Administration | Tablet Administration
Number analyzed (Participants) | 2000 | 2000
Sensitivity | 0.71 [.63 to .79] | .70 [.62 to .77]
Statistical Analysis 1: Comparison: Interviewer Administration; Each administration approach (interviewer and tablet) were separately tested against the reference measure; Test type: Other — Concurrent validity of the interviewer and self-administered versions of the TAPS Tool compared to the reference standard was assessed for Cannabis Use Disorder using receiver operator characteristic (ROC) curves; Sensitivity = .71, 95% CI 2-sided [.63 to .79]
Statistical Analysis 2: Comparison: Tablet Administration; Each administration approach (interviewer and tablet) were separately tested against the reference measure; Test type: Other — [test comment as in outcome 2, analysis 1]; Sensitivity = .70, 95% CI 2-sided [.62 to .77]

3. Primary Outcome: Diagnostic and Statistical Manual-5 (DSM-5) Cocaine and Amphetamine (Stimulant) Use Disorder Diagnosis Measured by the Modified World Mental Health Composite International Diagnostic Interview
Description: as for outcome 1
Time Frame: Baseline
Population: Adult primary care patients
Measure: Number (95% Confidence Interval); unit: Sensitivity
Arm/Group | Interviewer Administration | Tablet Administration
Number analyzed (Participants) | 2000 | 2000
Sensitivity | .57 [.47 to .67] | .60 [.50 to .69]
Statistical Analysis 1: Comparison: Interviewer Administration; Each administration approach (interviewer and tablet) were tested separately against the reference measure; Test type: Other — Concurrent validity of the interviewer and self-administered versions of the TAPS Tool compared to the reference standard was assessed for Cocaine and Amphetamine (Stimulant) Disorder using receiver operator characteristic (ROC) curves; Sensitivity = .57, 95% CI 2-sided [.47 to .67]
Statistical Analysis 2: Comparison: Tablet Administration; Each administration approach (interviewer and tablet) were separately tested against the reference measure; Test type: Other — Concurrent validity of the interviewer and self-administered versions of the TAPS Tool compared to the reference standard was assessed for Cocaine and Amphetamine (Stimulant) Use Disorder using receiver operator characteristic (ROC) curves; Sensitivity = .60, 95% CI 2-sided [.50 to .69]

4. Primary Outcome: Diagnostic and Statistical Manual DSM-5 Diagnosis of Heroin Use Disorder Measured by the The Modified World Mental Health Composite International Diagnostic Interview
Description: as for outcome 1
Time Frame: Baseline
Population: Adult primary care patients
Measure: Number (95% Confidence Interval); unit: Sensitivity
Groups:
- Tablet Administration: Tablet computer of a substance misuse screening instrument (TAPS Tool).
Arm/Group | Interviewer Administration | Tablet Administration
Number analyzed (Participants) | 2000 | 2000
Sensitivity | .66 [.53 to .77] | .66 [.53 to .77]
Statistical Analysis 1: Comparison: Interviewer Administration; Each administration approach (interviewer and tablet) were tested separately against the reference measure; Test type: Other — Concurrent validity of the interviewer and self-administered versions of the TAPS Tool compared to the reference standard was assessed for Heroin Use Disorder using receiver operator characteristic (ROC) curves; sensivity = .66, 95% CI 2-sided [.53 to .77]
Statistical Analysis 2: Comparison: Tablet Administration; Each administration approach (interviewer and tablet) were tested separately against the reference measure; Test type: Other — [test comment as in outcome 4, analysis 1]; Sensivity = .66, 95% CI 2-sided [.53 to .77]

5. Primary Outcome: Diagnostic and Statistical Manual DSM-5 Diagnosis of Tobacco Use Disorder Measured by the Modified World Mental Health Composite International Diagnostic Interview
Description: as for outcome 1
Time Frame: Baseline
Population: adult primary care patients
Measure: Number (95% Confidence Interval); unit: Sensivity
Arm/Group | Interviewer Administration | Tablet Administration
Number analyzed (Participants) | 2000 | 2000
Sensivity | .74 [.69 to .77] | .73 [.69 to .77]

6. Secondary Outcome: High Risk Tobacco Use Measured by the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST)
Description: The ASSIST assess lifetime and past 3 month substance use. A score on the Tobacco Scale from 0-3 is low risk, 4-26 is medium risk, and 27 or greater is high risk.The scales range is from 0 (no problem) to 31 (most severe problem).
Time Frame: Baseline
Population: Adult primary care patients
Measure: Number (95% Confidence Interval); unit: Sensitivity
Groups:
- Interviewer Administered: Interviewer administration of TAPS Tool. The ASSIST was interviewer administered as well.
- Tablet Administration: Tablet computer administration of TAPS Tool. The ASSIST was administered in by an interview.
Arm/Group | Interviewer Administered | Tablet Administration
Number analyzed (Participants) | 2000 | 2000
Sensitivity | .90 [.83 to .94] | .90 [.83 to .94]

7. Secondary Outcome: Unhealthy Cannabis Use
Description: The Time Line Follow Back Interview measures participant's self-reported number of days of cannabis use in the 30 days prior to the interview. Unhealthy cannabis use is considered 1 or more days of cannabis use in the past 30 days.The reported data represent the correlation between the TAPS Tool Cannabis Score and the Number of Days of cannabis use
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: Spearman Correlation
Groups:
- Interviewer Administered: Interviewer administered TAPS. The Time Line Follow Back was interviewer administered.
- Tablet Administration: Tablet computer administration of TAPS Tool. The TLFB was interviewer administered.
Arm/Group | Interviewer Administered | Tablet Administration
Number analyzed (Participants) | 2000 | 2000
Spearman Correlation | .85 [.82 to .88] | .84 [.81 to .88]

8. Secondary Outcome: Risky Alcohol Use
Description: Measured by the Alcohol Use Disorders Identification Test - Consumption Items. High risk on the AUDIT-C is 10 or higher. The higher the score on the AUDIT-C the greater the alcohol problem.The range of scores on the AUDIT-C is from 0 (no problem) to 12 (maximum problem).
Time Frame: Baseline
Population: Adult Primary Care Patients
Measure: Number (95% Confidence Interval); unit: Spearman Correlation
Groups:
- Self-administered: Self-administered TAPS Tool. The AUDIT-C was interviewer administered.
- Interviewer Administered: Interviewer administered TAPS Tool. The AUDIT-C was interviewer administered for both group
Arm/Group | Self-administered | Interviewer Administered
Number analyzed (Participants) | 2000 | 2000
Spearman Correlation | .63 [.59 to .66] | .64 [.61 to .68]
Statistical Analysis 1: Comparison: Self-administered; Each administration approach (interviewer and tablet) were tested separately against the reference measure; Test type: Other — The association on the interviewer and tablet computer administered versions of the TAPS Tool compared to the reference standard AUDIT-C score was assessed using Spearman Correlation; Spearman Correlation = .63, 95% CI 2-sided [.59 to .66] — The estimated value is a Spearman Correlation point estimate between TAPS Tool Alcohol Score and the AUDIT-C score. A Confidence Interval rather than a dispersion value is therefore reported
Statistical Analysis 2: Comparison: Interviewer Administered; Each administration approach (interviewer and tablet) was tested separately against the reference measure; Test type: Other — The association on the interviewer and tablet administered versions of the TAPS Tool compared to the reference standard of the AUDIT C score was assessed using Spearman Correlation; Spearman Correlation = .64, 95% CI 2-sided [.61 to .68] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Cigarette Smoking Risk
Description: Measured by the Fagerstrom Test for Nicotine Dependence. The range of scores on the Fagerstrom Test if from 0 (no risk) to 10 (highest risk). High risk is considered a score of 6 or greater.
Time Frame: baseline
Population: Adult Primary Care patients
Measure: Number (95% Confidence Interval); unit: Spearman Correlation
Groups:
- Self-administered TAPS Tool: Self-administered TAPS Tool. The Fagerstrom Test for Nicotine Dependence was administered by interviewer.
- Interviewer Administered: Interviewer administered TAPS Tool. The Fagerstrom Test was interviewer administered.
Arm/Group | Self-administered TAPS Tool | Interviewer Administered
Number analyzed (Participants) | 2000 | 2000
Spearman Correlation | .73 [.70 to .76] | .75 [.73 to .77]

10. Secondary Outcome: Smokeless Tobacco Questionnaire
Description: Any yes response to smokeless tobacco use reported on the smokeless tobacco questionnaire is considered high risk.
Time Frame: baseline
Population: Adult Primary Care patients
Measure: Number (95% Confidence Interval); unit: Spearman Correlation
Groups:
- Interviewer Administered: Interviewer administered TAPS Tool. The Smokeless Tobacco Questionnaire was interviewer administered.
- Self Administered: Self-administered TAPS Tool. The Smokeless Tobacco Questionnaire was interviewer administered.
Arm/Group | Interviewer Administered | Self Administered
Number analyzed (Participants) | 2000 | 2000
Spearman Correlation | .29 [.25 to .33] | .28 [.24 to .32]
Statistical Analysis 1: Comparison: Interviewer Administered; Each administration approach (interviewer and tablet computer) was tested separately against the reference measure; Test type: Other — The association on the interviewer and tablet computer administered versions of the TAPS Tool compared to the reference standard Smokeless Tobacco Questionnaire was assessed using Spearman Correlation; Spearman Correlation = .29, 95% CI 2-sided [.25 to .33] — The estimated value is a Spearman Correlation point estimate between the TAPS Tool Tobacco Score and the Smokeless Tobacco Questionnare. Confidence Interval rather than a dispersion value is therefore reported
Statistical Analysis 2: Comparison: Self Administered; Each administration approach (interviewer and tablet) were tested separately against the reference measure; Test type: Other; Spearman Correlation = .28, 95% CI 2-sided [.24 to .32] — The estimated value is a Spearman Correlation point estimate between TAPS Tool Tobacco Score and the score on the Smokeless Tobacco Questionnaire. A Confidence Interval rather than a dispersion value is therefore reported

11. Secondary Outcome: Cannabis Positive Oral Fluid Test
Description: Positive Oral Fluid Cannabis testing.
Time Frame: baseline
Population: Adult Primary Care Patients with oral fluid test results
Measure: Number; unit: Spearman Correlation
Groups:
- Interviewer Administered: Interviewer administered TAPS Tool. Oral Fluid Cannabis Test administered to the subset of participants that consented to provide an oral fluid sample. Oral fluid specimen was collected the same way in both arms.
- Self-administered TAPS Tool: Self administered TAPS Tool. Oral Fluid Cannabis Test administered to the subset of participants that consented to provide an oral fluid sample. Oral fluid specimen was collected the same way in both arms.
Arm/Group | Interviewer Administered | Self-administered TAPS Tool
Number analyzed (Participants) | 1802 | 1802
Spearman Correlation | .42 | .40
Statistical Analysis 1: Comparison: Interviewer Administered; Each administration approach (interviewer and tablet) were tested separately against the reference measure; Test type: Other — The association on the interviewer and tablet computer administered versions of the TAPS Tool compared to the reference standard of the results of the oral fluid test was assessed using Spearman Correlation; Spearman Correlation = .42, 95% CI 2-sided [.35 to .48] — The estimated value is a Spearman Correlation point estimate between TAPS Tool Cannabis Score and the results of the Oral Fluid Test. Confidence Interval rather than a dispersion value is therefore reported
Statistical Analysis 2: Comparison: Self-administered TAPS Tool; Test type: Other; Spearman Correlation = .40, 95% CI 2-sided [.33 to .46] — The estimated value is a point estimate of the Spearman Correlation between the TAPS Tool Cannabis Score and the Oral Fluid Cannabis Screen. A Confidence Interval rather than a dispersion value is therefore reported

ADVERSE EVENTS:
Time Frame: Baseline data only gathered in this study.
Description: The all cause mortality and serious adverse event data refer to the total combined sample (n = 2,000). We report the total sample here because all participants received both the interviewer and self-administered versions one immediately after the other in one single session.
Groups:
- All Participants: All participants enrolled in the study (because all participants were administered both the self-administered and the interviewer administered versions of the instrument, we are reporting adverse events for the total sample)
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/2000
Serious Adverse Events (participants affected / at risk) | 0/2000
Other Adverse Events (participants affected / at risk) | 16/2000
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=2000)
Blood on oral swab (Injury, poisoning and procedural complications) | 16 (16) — Traces of blood were seen on oral swab

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No